CLINICAL TRIAL: NCT01511315
Title: A Single-Center, Open-Label Study to Assess Change in Psychosocial and Occupational Dimensions With Ustekinumab Treatment of Moderate-to-Severe Psoriasis Evaluated With the Psychological General Well Being (PGWB), Work Productivity and Activity Impairment (WPAI), Psoriasis Quality of Life-12 Items (PQOL-12), and Dermatology Life Quality Index (DLQI)
Brief Title: The Quality of Life Study in Psoriasis Patients After Ustekinumab Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stelara QoL
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Psoriasis
Keywords: Moderate to severe psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ustekinumab (Experimental)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Biologic agent: sub-cutaneous injection at Weeks 0, 4, and then every 12 weeks thereafter.

SUMMARY:
This study aims to see if patient quality of life can be approved after treatment with an injectable medication called ustekinumab for the treatment of generalized psoriasis. The investigators hypothesize that the investigators will see improvement in quality of life.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate improvement in psoriasis patient quality of life after 36 weeks with ustekinumab through the use of validated dermatologic and non-dermatologic psychometric instruments.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are non-immunocompromised males or females 18 years of age or older
2. Subjects have moderate-to-severe (≥10% total body surface area) plaque psoriasis
3. Subject diagnosed at least 6 months prior to entering the study
4. Negative urine pregnancy test within 7 days before the first dose of ustekinumab in all women (except those surgically sterile or at least 5 years postmenopausal)
5. Sexually active subjects of childbearing potential must agree to use medically acceptable form of contraception during screening and throughout the study.
6. Are considered eligible according to the following tuberculosis (TB) screening criteria:

   * Have no history of latent or active TB prior to screening. An exception is made for subjects currently receiving treatment for latent TB with no evidence of active TB, or who have a history of latent TB and documentation of having completed appropriate treatment for latent TB within 3 years prior to the first administration of study agent. It is the responsibility of the investigator to verify the adequacy of previous antituberculous treatment and provide appropriate documentation.
   * Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
   * Have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study agent.
   * Within 1 month prior to the first administration of study agent, have a negative QuantiFERON-TB Gold test result, or have a newly identified positive QuantiFERON-TB Gold test result in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study agent. The QuantiFERON-TB Gold test are not required at screening for subjects with a history of latent TB and ongoing treatment for latent TB or documentation of having completed adequate treatment as described above; Subjects with documentation of having completed adequate treatment as described above are not required to initiate additional treatment for latent TB.
   * Have a chest radiograph both posterior-anterior and lateral views, taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current, active TB or old, inactive TB.
7. Subject meets concomitant medication requirements or agrees to complete a washout for restricted medications prior to starting the study.

   * Washout Period :

     * Must not have initiated or changed any other medications that could affect psoriasis (e.g. beta blockers, lithium salts, antimalarials) within the 4 week period prior to Week 0 or during the study
     * Subjects must not have received immunosuppressive, chemotherapy and/or systemic therapy including oral calcineurin inhibitors (such as cyclosporine), retinoids (Vitamin A and analogues), Methotrexate, Azathioprine, 6-thioguanine, Mycophenolate mofetil (MMF), Hydroxyurea, or cytokines (such as interferon-gamma) within the 4 week period prior to Week 0 or during the study
     * Subjects must not have received phototherapy (broadband or narrow-band UVB) within the 2 week period prior to Week 0 or during the study.
     * Subjects must not have received photochemotherapy (PUVA) within the 4 week period prior to week 0 or during the study
     * Subjects must not have received TNF-α inhibitors (such as infliximab, etanercept, adalimumab) within the 12 week period prior to Week 0 or during the study
     * Subjects must not have received alefacept within the 12 week period prior to Week 0 or during the study.
     * Subjects must not have received ustekinumab within the 12 week period prior to Week 0 or during the study.
     * Subjects must not have received treatment with an investigational drug within the previous 4 weeks or 5 half-lives prior to Week 0 (whichever is longer) or participation in another clinical trial within the 4 week period prior to Week 0 or during the study

Exclusion Criteria:

1. Subject is younger than 18 years of age.
2. Subject has less than 10% body surface involvement of his/her psoriasis.
3. Subjects with erythrodermic, pustular, or guttate psoriasis
4. History of known or suspected intolerance to any of the ingredients of the investigational study product.
5. Evidence of skin conditions other than psoriasis that would interfere with study-related evaluations of psoriasis.
6. Evidence of active infections such as fevers, chills, sweats, or history of untreated Lyme disease and active severe infections within 4 weeks before screening visit, or between the screening and Week 0 visits
7. Subject has a history of listeriosis, untreated TB, persistent or active infections requiring hospitalization or treatment with IV antibiotics, IV antiretrovirals, or IV antifungals within 30 days of baseline, or oral antibiotics, antivirals, or antifungals for purpose of treating infection, within 14 days of baseline.
8. Have a history of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, prior to screening.
9. Refer to inclusion criteria for information regarding eligibility with a history of latent TB.
10. Have had a Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening.
11. Have a chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of malignancy or current active infection, including TB.
12. Have had a nontuberculous mycobacterial infection or opportunistic infection (eg. Cytomegalovirus, pneumocystosis, aspergillosis) within 6 months prior to screening.
13. History of immune compromised status [e.g. human immunodeficiency virus (HIV) positive status or other immune suppressing drug] or a congenital or acquired immunodeficiency or subject testing positive for HIV, Hepatitis B, and/or Hepatitis C during screening procedures.
14. Subject has a poorly controlled medical condition including, but not limited to, unstable cardiovascular disease, poorly controlled diabetes, recent stroke, history of recurrent infections, or any other condition for which, in the opinion of the investigator, participation in the study would place the subject at risk
15. Subject has a history of or ongoing drug or alcohol abuse
16. Subject is not willing to comply with wash-out requirements (see above)
17. Subject is known, or suspected of being unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ustekinumab: Biologic agent: ustekinumab 45mg pre-filled syringes, subcutaneous injection at Weeks 0, 4, and then every 12 weeks thereafter. (each dose of 45mg for subjects weighing less than or equal to 100kg and 90mg for subjects weighing greater than 100kg)
Period: Overall Study
Arm/Group | Ustekinumab
Started | 36
Completed | 32
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Patients who did not complete the study (n=4) were not included in the baseline analysis.
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 41.2 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Quality of Life Measured by Change in Psychological General Well-Being Scale (PGWB) at Week 36 From Baseline.
Description: The PGWB is a self-administered validated psychometric instrument that measures a person's emotional well-being. It is specifically designed to be suitable for assessing psychological well being in the general medical population as opposed to a psychiatric population. The 22 questions of the PGWB can be further divided into 6 domains: anxiety, depressed mood, positive well being, self-control, general health, and vitality. The PGWB is graded on a Likert scale, which is commonly used in psychometric questionnaires where the answers range from strongly agree to strongly disagree with gradations in between. Total scores range from 0 to 110, with higher scores indicating better psychological well being. This instrument has been validated and used in many countries on large samples of the general population and on various subsets of medical patients.
Time Frame: Baseline, 36 weeks
Population: Only participants who completed the study were included in this analysis (n=32).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
units on a scale | 23.97 (3.65)

2. Secondary Outcome: Change in Psychological General Well-Being Scale (PGWB) Over Time (at Weeks 12 and 24) From Baseline
Description: as for outcome 1
Time Frame: Baseline, 12 and 24 weeks
Population: Only participants who completed the study were included in this analysis (n=32).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
units on a scale
  week 24 | 19.97 (3.93)
  week 12 | 18.63 (3.22)

3. Secondary Outcome: Change in Work Productivity and Activity Impairment Scale (WPAI-PSO) Over Time at Week 36 From Baseline
Description: The WPAI is a patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to general health or a specific health problem. The WPAI:PSO was created specifically for administering to patients with psoriasis. WPAI surveys were analyzed based on published algorithms to determine the following: current employment status, absenteeism (percentage of time missed from work due to psoriasis), presenteeism (percentage reduced productivity at work due to psoriasis), total activity impairment (TAI, percentage impairment in activities other than work due to psoriasis), and total work productivity impairment (TWPI, total percentage of work impairment from both absenteeism and presenteeism due to psoriasis). Each WPAI score is expressed as impairment percentages (0-100), with higher scores representing greater impairment (worse outcomes)
Time Frame: Baseline, 36 Weeks
Population: Only participants who completed the study were included in this analysis (n=32).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
units on a scale
  Employment | 1 (3.1)
  total work productivity impairment | -21.6 (36.4)
  Absenteeism | -4.8 (11.7)
  Presenteeism | 18.6 (35.2)
  total activity impairment | -26.6 (35.9)

4. Secondary Outcome: Change in Psoriasis Quality of Life - 12 Items (PQOL-12) Over Time (at Weeks 12, 24, and 36) From Baseline
Description: The PQOL-12 is a 12-item psoriasis-specific validated PRO based entirely on the patient's own assessment of their situation. The items were data-derived based on a series of population-based statistical studies and clinical trials conducted over a decade. The KMPI is one of the first tools used in dermatology to incorporate a validated PRO in critical medical decision-making. The scores range from 0-120 with higher scores indicating worse outcomes.
Time Frame: Baseline, 12, 24, and 36 Weeks
Population: Only participants who completed the study were included in this analysis (n=32).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
units on a scale
  week 36 | -38.34 (7.67)
  week 24 | -43.78 (8.01)
  week 12 | -40.06 (6.82)

5. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Over Time (at Weeks 12, 24, and 36) From Baseline
Description: The DLQI is a 10-item self-reported survey, which addresses feelings, daily activities, leisure, work, school, personal relationships, and treatment. Each question item is worth 3 points (total maximum score of 30), with higher score representing greater QoL impairment.
Time Frame: Baseline, 12, 24, and 36 Weeks
Population: Only participants who completed the study were included in this analysis (n=32).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
units on a scale
  week 36 | 12.91 (1.30)
  week 24 | 13.65 (1.23)
  week 12 | 13.00 (1.23)

6. Secondary Outcome: Percentage of Patients Achieving PGA of Clear or Almost Clear at Weeks 12, 24, and 36
Description: The Physician Global Assessment (PGA) scoring system is used to assess the severity and extent of psoriasis using a score of 0-6 (clear, almost clear, minimal, moderate, severe, to very severe) averaged over all lesions.
Time Frame: Weeks 12, 24, and 36
Population: Only participants who completed the study were included in this analysis (n=32).
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
percentage of participants
  week 36 | 71.8
  week 24 | 67.7
  week 12 | 56.3

7. Secondary Outcome: Percentage of Patients Achieving PASI-75 at Weeks 12, 24, and 36
Description: The Psoriasis Area and Severity Index (PASI) incorporates erythema, induration, and scale on a score of 0-4 weighted by percentage of body surface area involvement. PASI scores range from 0 to 72, with higher scores indicating worse disease. The percentage of patients achieving 75% reduction or better from the baseline PASI score in a designated time period has become the gold standard to measure the efficacy of psoriasis treatment options.
Time Frame: Weeks 12, 24, and 36
Population: Only participants who completed the study were included in this analysis (n=32).
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab
Number analyzed (Participants) | 32
percentage of participants
  week 36 | 78.1
  week 24 | 78.1
  week 12 | 71.9

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Ustekinumab
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No